CLINICAL TRIAL: NCT04683458
Title: GermanVasc/MDEpiNet Paclitaxel Study
Brief Title: Analysis of Linked Health Insurance Claims and Clinical Registries to Determine Device Surveillance With Paclitaxel-coated Medical Devices
Acronym: PacliVasc
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: GermanVasc (Other); BARMER (Other); MDEpiNet Verband Deutschland e.V. (Unknown)
Responsible Party: Principal Investigator, Christian Behrendt, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 20GermanVasc
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Paclitaxel Adverse Reaction; Outcome, Fatal
Keywords: Paclitaxel; Health Insurance Claims; Real-World Data; Quality Improvement
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Paclitaxel-coated devices: Patients with symptomatic peripheral arterial occlusive disease or diabetic foot syndrome with chronic limb-threatening ischaemia who underwent endovascular revascularisation of the peripheral arteries in the lower limbs with any drug-coated medical device (e.g., drug-eluting stent, drug-coated balloon).
  Interventions: Device: Drug-coated device
- Controlls: Patients with symptomatic peripheral arterial occlusive disease or diabetic foot syndrome with chronic limb-threatening ischaemia who underwent endovascular revascularisation of the peripheral arteries in the lower limbs with any medical device except drug-coated techniques (e.g., drug-eluting stent, drug-coated balloon).

INTERVENTIONS:
Device: Drug-coated device — The endovascular (intraluminal) application of a medical-device that was coated with paclitaxel
  Other Names: Drug-coated balloon; Drug-eluting stent; Paclitaxel-coated device; Paclitaxel-coated balloon; Paclitaxel-eluting stent; DES; DCB
  Groups: Paclitaxel-coated devices

SUMMARY:
The GermanVasc/MDEpiNet Paclitaxel Study, aims to use routinely collected data from health insurance claims and registries. The longitudinal data of Germany's second-largest insurance fund, BARMER, includes the outpatient and inpatient medical care provided to ≈9.4 million German citizens (13.2% of Germany's population) involving >21 million hospitalizations between January 1, 2008, and December 31, 2018. The BARMER cohort is similar to Western European countries and has been widely used for research projects. A regular random sample validation of internal and external validity is performed by the Medical Service of the Health Funds in Germany, and various peer-reviewed validation studies have been previously published. The GermanVasc clinical registry was implemented in 2018 as EU General Data Protection Regulation (GDPR) compliant registry platform to process routinely collected clinical data from more than 35 high-volume vascular centers in Germany. In an ongoing project of a large multispecialty and multidisciplinary research consortium (RABATT study, Principal Investigator: PD Dr. Christian-Alexander Behrendt), active surveillance and medical device evaluation methods were developed. The current study aims to determine the long-term safety and efficacy of paclitaxel-coated balloons and stents in peripheral arteries. It further aims to illuminate the underlying differences between the cohorts in randomized controlled trials (RCT) and real-world data that can possibly explain the diametrically opposed results in an ongoing international controversy.

ELIGIBILITY:
Inclusion Criteria:

* Fontaine stage II-IV
* Diabetic foot syndrome with chronic limb-threatening ischaemia
* Endovascular revascularisation procedure in the lower limbs
* Treatment between 2013 and 2017

Exclusion Criteria:

* Hybrid surgery
* Previous major amputation
* Previous cancer diagnosis
* Previous paclitaxel-exposure
* Previous percutaneous coronary intervention
* Previous revascularisation of the arteries in the lower limbs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 39 years who underwent first (index) endovascular revascularisation for symptomatic peripheral arterial occlusive disease or diabetic foot syndrome with chronic limb-threatening ischaemia in Germany between 2013 and 2017.
Sampling Method: Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality after 5-years | 5-years
Composite of all-cause mortality, myocardial infarction, and stroke after 5-years | 5-years
Composite of all-cause mortality and major amputation of the lower extremities after 5-years | 5-years
Target limb revascularization after 5-years | 5-years

SECONDARY OUTCOMES:
Incident cancer after 5-years | 5-years
Minor amputation of the target limb after 5-years | 5-years
Major amputation of the target limb after 5-years | 5-years
Rate of optimal pharmacological treatment with antithrombotics, antihypertensives, and lipid-lowering drugs | 1-year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of the responsible research group — http://germanvasc.de
- See also: Publication List of the Principal Investigator — http://christianbehrendt.net
- See also: Website of the German chapter of the Medical Device Epidemiology Network — http://mdepinet.de
- See also: Website of the US Center of the Medical Device Epidemiology Network — http://mdepinet.org